CLINICAL TRIAL: NCT03523988
Title: Effects of Pre-emptive Use of Combined Ibuprofen and Acetaminophen on Pain Control in Orthodontic Treatment
Brief Title: Pre-emptive Analgesics in Orthodontic Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Andrew Keith, Principal Investigator, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00001679
Record Dates: First submitted 2018-04-19; First posted 2018-05-14 (Actual); Results first posted 2018-10-30 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: NSAID; Pain Management
Keywords: Pre-emptive analgesics; Acetaminophen; Ibuprofen
MeSH Terms: conditions — Agnosia | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Intervention Model Description: Patients of the University of Washington Graduate Orthodontics Clinic
Who Masked: Participant, Care Provider, Investigator
Masking Description: The medications were prepared by the Kelley-Ross Compounding Group (Seattle, WA) and were identical in appearance. The bottles were labeled as "A", "B", or "C" and the identity of the medications were not revealed until after the data analysis was completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Acetaminophen (Active Comparator): Acetaminophen 650mg powder in gel capsule taken by mouth before entering appointment
  Interventions: Drug: Acetaminophen
- Ibuprofen (Active Comparator): Ibuprofen 400mg powder in gel capsule taken by mouth before entering appointment
  Interventions: Drug: Ibuprofen
- Acetaminophen and Ibuprofen (Experimental): Acetaminophen 650mg and Ibuprofen 400mg powder in gel capsule taken by mouth before entering appointment
  Interventions: Drug: Acetaminophen; Drug: Ibuprofen

INTERVENTIONS:
Drug: Acetaminophen — Acetaminophen gel capsule
  Other Names: Tylenol; Paracetamol
  Arms: Acetaminophen; Acetaminophen and Ibuprofen
Drug: Ibuprofen — Ibuprofen gel capsule
  Other Names: Advil
  Arms: Acetaminophen and Ibuprofen; Ibuprofen

SUMMARY:
This study is designed to determine if the preemptive use of a combination of acetaminophen and ibuprofen is more effective in reducing pain following orthodontic tooth movement when compared to the use of acetaminophen and ibuprofen alone.

DETAILED DESCRIPTION:
This study is designed to determine if the preemptive use of a combination of acetaminophen and ibuprofen is more effective in reducing pain following orthodontic tooth movement when compared to the use of acetaminophen and ibuprofen alone. Before their orthodontic appointment, participants will be administered acetaminophen (650mg), ibuprofen (400mg), or acetaminophen (650mg) + ibuprofen (400mg). Participants will be asked to record their pain intensity using a numerical (0-10) visual analog scale (VAS) during rest, light biting, and while chewing paraffin wax during the following time intervals: immediately following drug administration, 6 hours after, the morning after, and the second morning after orthodontic treatment.

ELIGIBILITY:
Inclusion Criteria:

-Orthodontic patient presenting for orthodontic treatment

Exclusion Criteria:

* History of taking an analgesic in the past six hours
* Hypersensitivity to ibuprofen or acetaminophen
* Aspirin-sensitive asthma
* Renal or liver impairment
* History of GI bleeding or ulcers
* Cardiovascular disease, recent myocardial infarction, heart failure, or coronary artery bypass graft surgery
* Currently taking antibiotics or other medications for a chronic systemic disease
* Bleeding disorder
* Pregnant or nursing

Ages: 12 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 73 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2017-06-23 (Actual); Study Completion 2017-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Marie Bollen, DDS, MS, PhD, Study Director — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Orthodontic patients that presented to the University of Washington Graduate Orthodontics Clinic between May 2nd and June 23rd, 2017 were approached for recruitment.
Pre-assignment Details: Participants were screened against a set of inclusion criteria during the informed consent process. If one or more of the inclusion were not met then the patient was not assigned to a group.
Period: Overall Study
Arm/Group | Acetaminophen | Ibuprofen | Acetaminophen and Ibuprofen
Started | 24 | 24 | 25
Completed | 7 | 8 | 7
Not Completed | 17 | 16 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acetaminophen | Ibuprofen | Acetaminophen and Ibuprofen | Total
Number analyzed (Participants) | 7 | 8 | 7 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.7 (9.6) | 25.9 (18.0) | 21.4 (15.3) | 23.1 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 3 | 12
  Male | 1 | 5 | 4 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 7 | 22

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS) Pain Scores at 6 Hours After Treatment
Description: Pain scores were measured and recorded by selecting a number [0-10] using a visual analog scale to assess pain during the following actions: jaw at rest, lightly biting, and chewing paraffin wax.
  The VAS consisted of a 10cm numerical scale from 0, representing "no pain," to 10, representing "worst possible, unbearable, excruciating pain."
Time Frame: 6 hours after orthodontic treatment
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Acetaminophen | Ibuprofen | Acetaminophen and Ibuprofen
Number analyzed (Participants) | 7 | 8 | 7
scores on a scale
  Rest | 0.6 (0.8) | 2.6 (2.2) | 1.0 (1.0)
  Biting | 2.0 (1.4) | 2.9 (2.5) | 2.0 (1.9)
  Chewing | 2.3 (1.4) | 4.0 (3.1) | 3.1 (2.5)
Statistical Analysis 1: Comparison: Acetaminophen vs Ibuprofen vs Acetaminophen and Ibuprofen; Test type: Superiority; p = 0.04, ANOVA — P-value for pain scores among the three comparison groups with jaw at rest
Statistical Analysis 2: Comparison: Acetaminophen vs Ibuprofen vs Acetaminophen and Ibuprofen; Test type: Superiority; p = 0.63, ANOVA — P-value for pain scores among the three comparison groups while lightly biting
Statistical Analysis 3: Comparison: Acetaminophen vs Ibuprofen vs Acetaminophen and Ibuprofen; Test type: Superiority; p = 0.41, ANOVA — P-value for pain scores among the three comparison groups while chewing paraffin wax

2. Primary Outcome: Visual Analog Scale (VAS) Pain Scores at 1 Day After Treatment
Description: as for outcome 1
Time Frame: 1 day after orthodontic treatment
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Acetaminophen | Ibuprofen | Acetaminophen and Ibuprofen
Number analyzed (Participants) | 7 | 8 | 7
scores on a scale
  Rest | 1.9 (2.5) | 2.0 (1.7) | 1.1 (1.2)
  Biting | 2.9 (2.5) | 2.5 (2.1) | 2.1 (2.7)
  Chewing | 3.6 (2.8) | 3.9 (3.1) | 2.7 (1.7)
Statistical Analysis 1: Comparison: Acetaminophen vs Ibuprofen vs Acetaminophen and Ibuprofen; Test type: Superiority; p = 0.65, ANOVA — P-value for pain scores among the three comparison groups with jaw at rest
Statistical Analysis 2: Comparison: Acetaminophen vs Ibuprofen vs Acetaminophen and Ibuprofen; Test type: Superiority; p = 0.82, ANOVA — P-value for pain scores among the three comparison groups while lightly biting
Statistical Analysis 3: Comparison: Acetaminophen vs Ibuprofen vs Acetaminophen and Ibuprofen; Test type: Superiority; p = 0.69, ANOVA — P-value for pain scores among the three comparison groups while chewing paraffin wax

3. Primary Outcome: Visual Analog Scale (VAS) Pain Scores at 2 Days After Treatment
Description: as for outcome 1
Time Frame: 2 days after orthodontic treatment
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Acetaminophen | Ibuprofen | Acetaminophen and Ibuprofen
Number analyzed (Participants) | 7 | 8 | 7
scores on a scale
  Rest | 1.3 (2.6) | 1.4 (1.5) | 0.4 (0.5)
  Biting | 2.3 (2.9) | 2.3 (1.5) | 0.9 (1.1)
  Chewing | 2.9 (2.9) | 3.1 (2.0) | 1.6 (1.4)
Statistical Analysis 1: Comparison: Acetaminophen vs Ibuprofen vs Acetaminophen and Ibuprofen; Test type: Superiority; p = 0.53, ANOVA — P-value for pain scores among the three comparison groups with jaw at rest
Statistical Analysis 2: Comparison: Acetaminophen vs Ibuprofen vs Acetaminophen and Ibuprofen; Test type: Superiority; p = 0.31, ANOVA — P-value for pain scores among the three comparison groups while lightly biting
Statistical Analysis 3: Comparison: Acetaminophen vs Ibuprofen vs Acetaminophen and Ibuprofen; Test type: Superiority; p = 0.37, ANOVA — P-value for pain scores among the three comparison groups while chewing paraffin wax

ADVERSE EVENTS:
Time Frame: Participants were given the contact information (phone and email) of the Lead Researcher to self-report any adverse events that occurred from the time they were administered their drug to the time of the last data entry (2 days following administration).
Arm/Group | Acetaminophen | Ibuprofen | Acetaminophen and Ibuprofen
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/25
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 1/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acetaminophen (N=24) | Ibuprofen (N=24) | Acetaminophen and Ibuprofen (N=25)
Acute Headache (General disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Low rate of participants returning results led to small number of participants analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2017-04-19): https://cdn.clinicaltrials.gov/large-docs/88/NCT03523988/Prot_003.pdf
  • Statistical Analysis Plan (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/88/NCT03523988/SAP_004.pdf
  • Informed Consent Form (2017-04-26): https://cdn.clinicaltrials.gov/large-docs/88/NCT03523988/ICF_005.pdf